CLINICAL TRIAL: NCT00191412
Title: Phase II Study of Single-Agent Alimta in the Treatment of Patients With Advanced and Metastatic Hepatoma
Brief Title: A Study of Pemetrexed in the Treatment of Patients With Advanced Metastatic Cancer of the Liver
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9417; H3E-US-S055
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-11-20 (Estimated); Status verified 2007-11

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms | interventions — Pemetrexed

INTERVENTIONS:
Drug: Pemetrexed

SUMMARY:
This study is to assess the response rate, toxicity, time-to-event efficacy, and potential markers of pemetrexed in patients with liver cancer.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cancer of the liver which is metastatic or locally recurrent and not amendable to curative therapy.
* Patient must have measurable disease
* Patient may have received prior arterial chemoembolization, completed 8 weeks prior to study enrollment, but no other previous chemotherapy
* Prior radiation is permitted, but must be completed at least 2 weeks prior to study enrollment.
* Prior central nervous system metastases are acceptable if the patient has received radiation ot the brain, is not on steroids, and does not have related symptoms.

Exclusion Criteria:

* Patients who have had prior therapy with Pemetrexed.
* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer, are excluded if there is any evidence of other malignancy being present within the last five years. Patients are also excluded if their previous cancer treatment contraindicates this protocol therapy.
* Patients who have received radiation to more than 25% of marrow

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41
Dates: Start 2005-01; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Antitumor activity as measured by Response Evaluation Criteria in Solid Tumors

SECONDARY OUTCOMES:
Toxicity measured by CTCAE grading
Duration of response: First complete or partial response until progressive disease (PD) or death of any cause
Duration of stable disease: Enrollment to PD or death of any cause
Time to treatment failure: Enroll. to PD, death of any cause, early discontinuation of treatment for any reason other than adequate response or start of new therapy
Progression-free survival: Enroll. to PD or death of any cause
Overall survival: Enroll. to death of any cause

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT) - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Denver, Colorado, United States

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com